CLINICAL TRIAL: NCT03588260
Title: Respiratory Muscle Strength in Patients With Idiopathic Pulmonary Fibrosis: The Relationship With Exercise Capacity, Physical Activity Level, and Quality of Life
Brief Title: Respiratory Muscle Strength in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Other Study IDs: IPF_MIP/MEP
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; respiratory muscle strength; physical activity; quality of life; dyspnea; fatigue severity; exercise capacity
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Motor Activity; Dyspnea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic pulmonary fibrosis: The patients who have agreed to participate in the study from patients diagnosed with idiopathic pulmonary fibrosis referred to the center of pulmonary rehabilitation from the interstitial lung disease polyclinic.
  Interventions: Other: no intervention - cross-sectional observational only
- Healthy subjects: The healthy adults without additional disease
  Interventions: Other: no intervention - cross-sectional observational only

INTERVENTIONS:
Other: no intervention - cross-sectional observational only — no intervention - cross-sectional observational only

SUMMARY:
Respiratory muscle strength, dyspnea perception, physical activity and quality of life measurements will be performed and groups will be compared in two groups consisting of patients with idiopathic pulmonary fibrosis referred to pulmonary rehabilitation clinic and healthy volunteers in similar age range.

DETAILED DESCRIPTION:
The patients who have agreed to participate in the study from patients diagnosed with idiopathic pulmonary fibrosis referred to the center of pulmonary rehabilitation from the interstitial lung disease polyclinic will be included in the study. In addition, a healthy adult control group will be established from similar age groups. The two groups will be compared in terms of outcome measures.The study outcome measurements are maximum inspiratory/expiratory muscle strength , international physical activity questionaire, modified Medical Research Council dyspnea scale, Short form 36 quality of lide questionaire, fatigue severity scale, six minute walking test.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70
* Patients signing informed consent form
* Patients diagnosed with idiopathic pulmonary fibrosis.

Exclusion Criteria:

* Patients who use steroids for less than 1 year
* The patient does not want to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who have agreed to participate in the study from patients diagnosed with idiopathic pulmonary fibrosis referred to the center of pulmonary rehabilitation from the interstitial lung disease polyclinic will be included in the study. In addition, a healthy adult control group will be established from similar age groups. The two groups will be compared in terms of outcome measures.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory muscle pressure | 15 minutes
  The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Maximum expiratory muscle pressure | 15 minutes
  The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
The distance covered in six-minute walk test | 10 minutes
  The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Patients were told that they should walk as fast as they can walk. Before and after the test, oxygen saturation, heart rate, Borg fatigue rating, and walking distance were recorded.
International Physical Activity Questionnaire | 15 minutes
  The International Physical Activity Questionnaire (IPAQ) was developed as an instrument for cross-national monitoring of physical activity and inactivity. This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
The Quality of Life Questionaire | 20 minutes
  Short Form 36

SECONDARY OUTCOMES:
The modified Medical Research Council (mMRC) scale | 3 minutes
  Dyspnea perceptions during daily life activities will assess according to the modified Medical Research Council (mMRC) scale. The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "0" means no dyspnea perception, "4" means severe dyspnea perception.
The fatigue severity scale | 15 minutes
  * A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity.
  * The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree
  * The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity
  * Another way of scoring: mean of all the scores with minimum score being 1 and maximum score being 7
  * Self-report scale

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)